CLINICAL TRIAL: NCT04240691
Title: Instacare: A Prospective Study of Clinical Outcomes Following Rapid ART Initiation Among Persons With HIV and Out of Care
Brief Title: Instacare - Rapid ART Initiation Among Persons With HIV and Out of Care
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Susan Little, MD, Professor, University of California, San Diego
Other Study IDs: 191875
Record Dates: First submitted 2020-01-14; First posted 2020-01-27 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Hiv; HIV Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stored Samples Containing DNA: blood and cells containing genetic materials will be stored. The blood and cells will be identified only be an identification number. However, there is an inherent risk of inadvertent disclosure of identity because DNA can be used to identify an individual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 60-Minutes-For-Health: 60-Minutes-for Health: this is a psychological intervention which seeks to correct factors underlying decisions to delay or avoid HIV care and strengthen abilities to overcome HIV care utilization barriers. This is achieved through assistance identifying and reducing misinformation guiding HIV care attendance decisions; enhancing motivation to maintain HIV care via personal health goals; building skills for coping with negative feelings related to living with HIV; and increasing self-efficacy for navigating structural barriers and maintaining HIV care amidst competing priorities.
  Interventions: Behavioral: 60-Minutes-For-Health
- Time-and-Attention Control Session: 60 Minute diet & nutrition control session
  Interventions: Other: Time-and-Attention Control Session

INTERVENTIONS:
Behavioral: 60-Minutes-For-Health — Refer to description under Groups
  Groups: 60-Minutes-For-Health
Other: Time-and-Attention Control Session — Refer to description under Groups
  Groups: Time-and-Attention Control Session

SUMMARY:
This study aims to evaluate two ways to help people re-engage with healthcare. The first is to assess if providing HIV treatment on the first visit (or within 1 week) can help people re-engage with care and ultimately stay in care after 24 and 48 weeks. It will also assess the success of starting treatment immediately by measuring the HIV virus in people's bloodstream after 24 and 48 weeks.

The second part of this study is to assess a new behavioral treatment called 60-Minutes-for-Health which aims to help people identify and overcome barriers to HIV care, to help with motivation maintaining in care, to help cope with negative feelings about HIV, and to help increase self-reliance in seeking healthcare amid other things that are happening in your life.

DETAILED DESCRIPTION:
The human immunodeficiency virus (HIV) continues to cause significant illness and death in the USA despite availability of effective treatment. People who are aware of their HIV status, but who are out of care and not on medications, are therefore at risk of developing HIV related health problems. In addition, people with HIV who are out of care are at greater risk of transmitting HIV compared to people on HIV treatment with suppressed levels of virus in plasma. To date, there are no interventions that have been shown to successfully link this "out of care" population back into care and successfully maintain viral suppression.

This study will test a strategy of providing immediate HIV therapy drugs, linkage to care, and a randomized intervention (60-minutes for health or diet and nutrition session). The goal of the study is to demonstrate that the 60-Minutes-for-Health intervention improves the rate of viral suppression at 24 weeks.

The use of rapid antiretroviral therapy (rapid ART), defined as the initiation of ART within 7 days of HIV diagnosis, has been associated with improved rates of linkage to care, retention in care and virological suppression after 1 year among persons newly diagnoses with HIV. In addition, the behavioral intervention, "60-Minutes-for-Health", was shown in a pilot study to improve retention in care among PWH-OOC. We aim to undertake a study to evaluate the feasibility of providing rapid-ART to people who are aware of their HIV status, but have been out of care at the time they re-engage in care. In addition, study participants will be randomized to either the "60-Minutes-for-Health" intervention or a 60 minute diet and nutrition control session.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Documented HIV infection status (or rapid HIV will be repeated);
* Out-of-care defined as not seen in HIV provider clinic for ≥6 months AND not receiving ART for ≥1 month (by self-report);
* Available for follow-up according to schedule of evaluations.

Exclusion Criteria:

* Co-morbid condition(s) that in the opinion of the investigator could limit the participant's ability to comply with the visit schedule or safely initiate rapid ART (e.g. psychiatric comorbidities or suspected central nervous system opportunistic infection);
* Prior ART regimens that in the opinion of the investigator precludes selection of a treatment option likely to result in virologic suppression (e.g. documented treatment failure on INSTI based regimen and multiple prior NRTI, NNRTI and PI regimens or documented resistance mutations likely to result in treatment failure)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Potential subjects from UCSD Owen Clinic that fulfill the entry criteria will be contacted and offered an appointment for study recruitment
  2. Subjects identified in the UCSD emergency department HIV screening program will be contacted and offered an appointment for study recruitment
  3. San Diego Public Health Department (SDPHD) has implemented routine evaluations of their local HIV surveillance data in conjunction with other data to identify PWH who may be OOC33. This Data to Care program results in the evaluation of ~ 250 new cases per year in San Diego (~20-21 PWH-OOC a month), many of whom are found to be viremic and out-of-care. Once located, SDPHD will offer immediate transportation vouchers (Lyft) to and from the AVRC to expedite study enrollment and rapid ART start.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Viral Suppression | Week 24
  HIV VL ≤50 at week 24
Retention in Care | Week 24
  Two clinical care visits between enrollment and week 24 at least 90 days apart

SECONDARY OUTCOMES:
ART Initiation | Week 4
  The self-reported initiation of ART
Viral Suppression | Week 48
  The proportion of participants with HIV VL ≤50 at week 48
Retention in care | Week 48
  The proportion of participants with ≥2 clinical care visits >90 days apart between enrollment and week 48
Genotypic susceptibility score comparison | Week 24 and 48
  To compare discrete genoptypic susceptibility score (derived from banked archive genotype at enrolment) between individuals with and without virologic suppression at week 24 and 48
Rapid ART acceptability | Week 4-8
  ACASI-delivered survey items administered to all participants.Responses are given on a 5-point Likert-type scale and recoded so that more favorable assessments are reflected in higher ratings (1=Least favorable, 5=Most favorable).A mean composite score will be created for sub-scales with ≥3-items. Mean scores for the seven acceptability metrics below will be computed for the total sample and each study arm (intervention, control).Among a subset of participants enrolled in four focus groups (10 participants each) will be held. Our interview guide will elicit feedback on the seven theory-based acceptability/feasibility metrics:affective attitudes towards rapid ART,perceived burden or reasons for discontinuation/dropout, perceived effectiveness, potential consequences (ethical, unintended, or side-effects) of rapid ART,willingness to participate in rapid ART,perceived costs (financial,social,emotional,physical) of rapid ART,perceived user experiences and satisfaction with rapid ART.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Little, MD, Principal Investigator — UC San Diego AntiViral Research Center (AVRC)
Locations (2):
- United States (2):
  - UC San Diego AntiViral Research Center (AVRC), San Diego, California
  - UC San Diego Owen Clinic, San Diego, California

IPD SHARING:
Plan to Share IPD: Undecided
Collaboration with other Academic Research Groups studying Rapid ART: Coded data, that have been stripped of identifiers, from HIV infected participants may be shared with research investigators in the U.S. and abroad, to better understand the acceptability and durability of Rapid ART and to gain a better understanding of this treatment strategy in all populations. InstaCare investigators will maintain the code book in order to access identifiers to link data sets outside of the InstaCare research study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT04240691/Prot_SAP_000.pdf